CLINICAL TRIAL: NCT00136396
Title: An Open Label, Phase I/II Trial of Rituximab Therapy for Steroid-Refractory Chronic Graft vs. Host Disease
Brief Title: Rituximab Therapy for Steroid-Refractory Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-120
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Graft vs Host Disease
Keywords: Steroid-refractory Chronic Graft vs. Host Disease; Chronic Graft vs. Host Disease; GVHD; steroid-refractory; rituximab
MeSH Terms: conditions — Graft vs Host Disease | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — Given once weekly for 4 weeks followed by a 4 week observation therapy.

SUMMARY:
The purpose of this study is to determine if rituximab is a safe and effective therapy for steroid-refractory chronic graft versus host disease (GVHD).

DETAILED DESCRIPTION:
Patients will receive rituximab intravenously one time per week for four consecutive weeks. Once therapy is completed, the patient will have weekly visits with their physician for four more weeks, at which they will complete a simple questionnaire designed to evaluate the severity of chronic graft versus host disease.

At the end of the eighth week on the study (4 weeks of study treatment and 4 weeks of observation), patients will be evaluated to determine whether their chronic graft versus host disease (GVHD) has resolved.

If chronic graft versus host disease has resolved entirely, the patient will be monitored for the remainder of the year.

If after the initial eight weeks on the study the patient still has symptoms or signs of GVHD, they may receive a second four week study treatment.

If the patients' chronic GVHD reappears after receiving either one or two courses of rituximab, a third and final four week course of medication can be given provided it has been at least eight weeks since the last dose.

Blood tests will be performed at the beginning of the study, after 8 weeks on the study, after 16 weeks on the study and at the end of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of matched related, matched unrelated, or mismatched stem cell transplantation
* At least 180 days since allogeneic stem cell transplantation procedure
* Patients must have steroid-refractory chronic GVHD, defined as having persistent signs and symptoms despite the use of prednisone
* Stable dose of corticosteroids for 4 weeks prior to enrollment
* Adequate bone marrow function: absolute neutrophil count (ANC) > 500/mm; platelets > 20,000 ul
* Adequate renal function: creatinine < 3.0 mg/dl
* Adequate hepatic function: bilirubin < 3.0 mg/dl; AST < 90 IU

Exclusion Criteria:

* Prednisone requirement greater than 2 mg/kg/day or equivalent
* Known life-threatening sensitivity to rituximab or other anti-B cell antibody.
* Prior exposure to any new immunosuppressive medication in the preceding 4 weeks prior to enrollment.
* Active, uncontrolled infection
* Evidence of natural exposure to hepatitis B or C.
* Active malignant disease relapse
* Donor lymphocyte infusion within the preceding 100 days.
* Life expectancy of less than 3 months.
* Pregnancy or lactation
* Evidence of HIV seropositivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of up to three four week courses of rituximab in steroid-refractory chronic GVHD | 2 years

SECONDARY OUTCOMES:
To determine the effects of rituximab therapy on quality of life of patients with steroid-refractory GVHD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Corey S. Cutler, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Cutler C, Miklos D, Kim HT, Treister N, Woo SB, Bienfang D, Klickstein LB, Levin J, Miller K, Reynolds C, Macdonell R, Pasek M, Lee SJ, Ho V, Soiffer R, Antin JH, Ritz J, Alyea E. Rituximab for steroid-refractory chronic graft-versus-host disease. Blood. 2006 Jul 15;108(2):756-62. doi: 10.1182/blood-2006-01-0233. Epub 2006 Mar 21. PMID 16551963